CLINICAL TRIAL: NCT01206673
Title: Evaluation of Macrophagic Activation and Immunophenotypic Profile of Patients With Gaucher's Disease.
Brief Title: Macrophagic Activation and Immunophenotypic Profile of Patients With Gaucher's Disease
Acronym: Gaucher
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09/07-I
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Patients With Gaucher's Disease
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood sampling — One blood sampling is required for the research

SUMMARY:
The aim of this study is to evaluate macrophaging activity and immunologic profile of patients with Gaucher 's disease. For this, one blood sampling will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age equal or above 18.
* Patients with Gaucher 's disease treated in the "Grand Ouest" competence center
* patients affiliated to social security
* Informed consent signed

Exclusion Criteria:

- Children (age<18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the implication of acquired and inherent immunity in the Gaucher's clinical phenotype at moment of blood sampling

SECONDARY OUTCOMES:
to find new activity mark for Gaucher's disease by studying macrophagic activation's markers.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nantes Hospital, Nantes
  - CHU of Rennes, Rennes